CLINICAL TRIAL: NCT02681107
Title: Accelerated Partial Breast Irradiation Using Five Daily Fractions: A Single Arm, Phase II, Prospective Cohort Study to Examine Cosmetic Outcomes and Toxicity (The ACCEL Trial)
Brief Title: APBI: 27Gy in 5 Fractions for Early Breast Cancer
Acronym: ACCEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-16-0006; No. 11629-27/5-01 (Other Grant/Funding Number: TBCC CTU)
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Radiation therapy; Accelerated partial breast irradiation (APBI); Breast conserving surgery; Stage 1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 2 - Irradiation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Single cohort to receive Accelerated Partial Breast Irradiation (APBI) 27Gy in 5 fractions
  Interventions: Radiation: APBI 27Gy in 5 fractions

INTERVENTIONS:
Radiation: APBI 27Gy in 5 fractions — Patients will be treated with 3-D conformal, external beam, partial breast RT to deliver 27 Gy in 5 daily fractions using 3-5 beams on a linear accelerator. The target PTV will be the CT-visible seroma plus a 1cm margin to form the CTV (minus 5mm from skin and excluding chest wall) and a further 7mm to form the PTV. Real time review will ensure compliance with target and normal tissues dose constraints in this multi-institutional study. Any (or no) systemic therapy is permitted.

SUMMARY:
This study will test the safety of partial breast RT using 27Gy in 5 daily fractions which is expected to be equally tolerated as standard whole breast irradiation (WBI) based on radiobiologic modeling of the fibrosis response of normal tissues but be more convenient and less costly than 3-6 weeks of standard WBI. 274 women will be treated. Rates of fibrosis and cosmesis at 2 years will be compared to data already collected using standard WBI in the Canadian RAPID trial.

DETAILED DESCRIPTION:
Background: Previously, accelerated partial breast irradiation (APBI) using 3D conformal external beam techniques to deliver 38.5Gy in 10, twice daily, fractions caused worse fibrosis and cosmetic deterioration than standard whole breast irradiation (WBI) following breast conserving surgery (BCS) for women with early breast cancer. Over the decade since the original APBI technique was designed, long-term outcomes of various breast RT fractionation regimens have become available and suggest that normal tissue fibrosis and cosmesis varies with the radiobiological constant: α/β=2 rather than α/β=3.4 as previously estimated. Radiobiologic modeling using α/β=2, indicates that a dose of 27Gy in 5 daily treatments should result in comparable late effects as 42.5Gy in 16, or 50Gy in 25 fractions. This clinical trial will validate the safety of a short, convenient and less costly APBI using 27Gy in 5 daily fractions.

Objective: To determine the cosmetic and normal tissue outcomes of APBI using 3D-conformal RT with 27Gy in 5 fractions over 1 week.

Methods: A single-arm, phase II, non-inferiority, prospective study will be conducted. 274 women with newly diagnosed, invasive or in-situ ductal carcinoma treated with BCS and sentinel lymph node biopsy (or axillary dissection) who are candidates for WBI alone, will be treated. Subjects will be age 50 years and older, with tumors less than 3cm diameter, with negative margins and nodes and with excellent or good baseline cosmetic outcome following BCS. Patients with extensive ductal carcinoma in-situ, BRCA mutations, Grade 3 cancers with lymphatic or vascular invasion, or lobular carcinoma will be excluded. These selection criteria are similar to the Canadian RAPID trial. In the first phase of the study, 150 patients will be recruited and interim analyses will be conducted to rule out unacceptable toxicity at 2 years.

Study endpoints: The primary endpoint will be the proportion of women who retain an Excellent or Good cosmetic score at 2 years using the EORTC Cosmetic Rating System and clinical photographs taken prior to, and at 1 and 2 years after RT. Secondary endpoints will include rates and grades of breast fibrosis, induration, telangiectasia, breast pain, ipsilateral breast tumor recurrence, overall and breast cancer-specific survival and subsequent mastectomy rates.

Sample size, statistical analyses: In the RAPID trial, 88% of patients with Excellent or Good cosmesis prior to RT had Excellent or Good scores at 3 years. Only patients with Excellent/Good cosmesis at baseline will be included in the current study. The proportion of women with Excellent/Good cosmesis at 1 and 2 years will be calculated. Using 80% power, a non-inferiority margin of 0.08 and a one-sided binomial test for non-inferiority and a significance level of 0.05, will require a sample size of 249 women with evaluable 2-yr cosmesis. 274 patients will be recruited to allow for a 10% drop-out rate. To ensure safety, a first interim analysis with Grade 2 or higher breast fibrosis as the primary endpoint, will be conducted when 50 patients have completed their 1-year assessment and repeated when 50 patients have completed their 2-year follow up. If the rate of Grade 2 or higher fibrosis exceeds 5% at either time point, trial accrual will be suspended.

Feasibility: Over 600 women eligible for this protocol receive RT in Alberta each year. If 30% accept study participation, accrual will be complete in <2 years.

ELIGIBILITY:
Inclusion Criteria:

* Female, with new invasive or in-situ ductal carcinoma of the breast
* Treated with Breast conserving surgery (BCS) with negative margins
* pN0 on sentinel node biopsy or axillary dissection; cN0 if DCIS alone
* Maximum pathologic tumor diameter is 3.0 cm (invasive or DCIS)
* No clinical or imaging evidence of distant metastases
* Age 50 years or older at diagnosis
* No contraindications to breast irradiation
* Excellent or Good overall cosmetic score at baseline following BCS
* Able and willing to provide written informed consent
* Available for 2 year follow up at the treating RT centre

Exclusion Criteria:

* Age < 50 years at diagnosis
* BRCA 1 or 2 pathogenic mutation
* Pathologic tumor diameter >3cm (including DCIS+invasive disease)
* Lobular histology alone
* Triple negative (ER-, PR-, HER2-) or HER2 overexpressing disease
* Margin (other than deep) <2 mm
* Presence of both Grade 3 and lymphatic or vascular invasion
* Fair or Poor overall cosmetic score at baseline following BCS
* Presence of ipsilateral breast implants
* Inability to develop an APBI plan meeting all dosimetry constraints
* Unable to start RT within 16 weeks of BCS or 8 weeks of last iv chemotherapy
* Unable or unwilling to sign informed consent document or attend for 2-year cosmetic assessment at the treating RT centre
* Potential contraindications for breast RT including a confirmed diagnosis of lupus, scleroderma, or pregnancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Excellent or Good Global cosmetic score | 2 years
  Global cosmetic score assessed by trained observers and patients themselves using the European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer rating system for cosmetic assessment; rate of deterioration from Excellent/Good to Fair Poor. This will be augmented by assessment of clinical photographs prior to and at 1 and 2 years after radiation therapy (RT).

SECONDARY OUTCOMES:
Breast induration | 2 years
  Radiation Therapy Oncology Group (RTOG) Late Radiation Morbidity Scoring Scheme, rate of Grade 2+ subcutaneous fibrosis
Breast pain | 2 years
  Patient reported average and worst pain in the treated breast over the week prior to assessment
Local recurrence | 2 and 5 years
  Any new invasive or in situ breast cancer within the ipsilateral breast

CONTACTS AND LOCATIONS:
Overall Officials: Petra Grendarova, MD, Principal Investigator — Tom Baker Cancer Centre, Alberta Health Services
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
At least one peer-review publication will be prepared by the investigators following the conclusion of the study. In addition, an abstract to report interim results following the 1-year, interim cosmetic evaluation may be submitted to the annual Canadian Association of Radiation Oncology and/or San Antonio Breast Cancer Symposium scientific meetings.
  Authorship will include the named investigators involved in the development of the grant proposal plus additional authors proportional to subject accrual, participation in the cosmetic photograph review panels and/or other contributions to study analysis or success.

REFERENCES:
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717